CLINICAL TRIAL: NCT06190275
Title: A Single-Arm Clinical Study of Autologous Tumor-Infiltrating Lymphocyte Infusion (GT201) in Combination With PD-1 Inhibitor for Advanced Head and Neck Tumors
Brief Title: Clinical Study of GT201 in Combination With PD-1 Inhibitor for Advanced Head and Neck Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-201-003
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT201 in combination with PD-1 inhibitors treatment group (Experimental)
  Interventions: Biological: GT201 in combination with PD-1 inhibitors

INTERVENTIONS:
Biological: GT201 in combination with PD-1 inhibitors — GT201 in combination with a PD-1 inhibitor for advanced head and neck tumors

SUMMARY:
This study is a single-arm early exploratory clinical study. designed to evaluate the safety and tolerability of GT201 in combination with a PD-1 inhibitor for the treatment of advanced head and neck tumor subjects with safety and tolerability, as well as pharmacokinetic characterization and efficacy The study consists of two phases.

The study consists of two phases, a dose-escalation phase and a dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily join the study, signed informed consent form,, willing and able to comply with the study protocol;
* 2. Age 18 to 70 years old;
* 3. Diagnosis with recurrent or metastatic head and neck malignant tumors and received≤2 lines of systemic therapy;
* 4. Have at least one measurable lesion that is untreated with radiotherapy or other local therapies, is accessible for tumor tissue collection (assessed by the investigator), and can provide a tissue block with a mass ≥1.0 g (approximately 1.5 cm in diameter) for autologous tumor-infiltrating lymphocyte (TIL) preparation. The tissue collection procedure should be minimally invasive whenever possible.
* 5. After tumor sampling, have at least one measurable lesion as defined by RECIST v1.1.
* 6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* 7. Expected survival time of ≥ 12 weeks;
* 8. Adequate function of major organs, with the following requirements (administration of any blood components or cell growth factors is not allowed within 14 days prior to surgery):

  1. Hematology:

     * Absolute Neutrophil Count (ANC) ≥ 1.0×10⁹/L;
     * Lymphocyte Count (LC) ≥ 0.5×10⁹/L;
     * Platelet Count (PLT) ≥ 80×10⁹/L;
     * Hemoglobin (Hb) ≥ 90 g/L.
  2. Liver function:

     * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and Alkaline Phosphatase (ALP) ≤ 2.5×Upper Limit of Normal (ULN);
     * Total Bilirubin (TBIL) ≤ 1.5×ULN.

     The following exceptions apply:
     * For confirmed liver metastases: AST and/or ALT ≤ 5×ULN;
     * For confirmed liver or bone metastases: ALP ≤ 5×ULN;
     * For confirmed Gilbert's syndrome: TBIL ≤ 3.0 mg/dL.
  3. Renal function:

     • Creatinine Clearance (CrCL) ≥ 45 mL/min (calculated by the Cockcroft-Gault formula), or serum creatinine within the normal range.
  4. Coagulation function:

     * Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN;
     * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5×ULN simultaneously.
  5. Adequate cardiac function.
  6. Adequate pulmonary function.
* 9. For women of childbearing potential who have not undergone surgical sterilization:

  * Agree to use at least one medically approved contraceptive method (e.g., intrauterine device, oral contraceptives, or condoms) during the study treatment period and for 1 year after the end of study treatment;
  * Serum human chorionic gonadotropin (HCG) test result must be negative at screening.
* 10. Adverse reactions caused by prior therapies have resolved to ≤ Grade 1 per CTCAE v5.0 before tumor sampling.
* 11. For subjects enrolled due to insufficient efficacy or intolerability of prior therapies, medical records documenting disease status after prior treatment or imaging records of lesion assessment must be available before tumor sampling.

Exclusion Criteria:

* 1. Uncontrolled local or systemic infections of the oral cavity, head, or neck; any active autoimmune disease, history of autoimmune disease, or disease requiring systemic corticosteroid therapy or immunosuppressive drugs (prednisone equivalent dose > 10 mg/day).
* 2. Subjects with uncontrollable tumor-related pain assessed by the investigator. Subjects requiring analgesic treatment must be on a stable analgesic regimen at study entry; symptomatic lesions eligible for palliative radiotherapy should have completed treatment prior to study entry.
* 3. Bleeding events occurring within 3 months prior to screening, including but not limited to gastrointestinal bleeding caused by fundic or esophageal varices, increased bleeding risk due to portal hypertension, active gastrointestinal bleeding, etc.; or subjects assessed by the investigator as having a high risk of major bleeding, including but not limited to tumors encasing or invading major blood vessels [i.e., carotid artery, jugular vein, bronchial artery] and/or exhibiting other high-risk features (e.g., fistula, significant cavitary lesions, history of bleeding [≤ 60 days from signing the ICF]).
* 4. Arterial/venous thrombotic events occurring within 6 months prior to screening, such as cerebrovascular accident, deep vein thrombosis, and pulmonary embolism.
* 5. A history of interstitial pneumonia, clinically significant active pneumonia at screening, or other respiratory diseases that severely impair pulmonary function.
* 6. A history of clinically significant cardiovascular disease, including but not limited to: (1) congestive heart failure (NYHA class > 2); (2) unstable angina pectoris; (3) myocardial infarction within the past 3 months; (4) any supraventricular or ventricular arrhythmia requiring treatment or intervention.
* 7. Subjects with ≥ 3 untreated central nervous system (CNS) metastases at screening. Exclusion exception: Subjects with ≤ 3 CNS metastases, with the largest lesion < 1 cm in diameter, no peritumoral edema on brain imaging (MRI or CT), and no evidence of progressive CNS disease on brain imaging for at least 3 months after treatment may be enrolled.
* 8. Ineligible for enrollment if spinal cord compression has not been relieved by surgery and/or radiotherapy. Exclusion exception: Subjects with active CNS metastases are excluded, except for those with stable brain metastases who have not required medical treatment for 3 months and are not dependent on corticosteroids.
* 9. A history of malignant tumors other than the target indication within 5 years prior to screening (excluding adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, and breast ductal carcinoma in situ after radical resection), unless the investigator determines that the benefits to the subject outweigh the risks.
* 10. Presence of refractory or intractable epilepsy, massive pleural effusion, ascites, pericardial effusion, etc., that cannot be controlled by medication, or contraindications to interleukin-2 (IL-2) use.
* 11. A history of infectious diseases within 1 year prior to screening, such as HIV, syphilis, active viral hepatitis, active pulmonary tuberculosis, active EBV and/or CMV infection; or a history of active pulmonary tuberculosis infection for more than 1 year without standard treatment. Active hepatitis B or hepatitis C is excluded. Enrollment exceptions:

  * Subjects positive for HBsAg or HBcAb may participate if HBV DNA test results are below the lower limit of normal (LLN) at the testing site;
  * Subjects positive for HCV antibody may participate if HCV RNA test results are below the LLN at the testing site.

Carriers enrolled in the study should receive antiviral therapy as appropriate and undergo regular nucleic acid copy number quantitative testing during the study period.

* 12. Use of anti-angiogenic agents (e.g., bevacizumab, a VEGF inhibitor) within 4 weeks prior to surgical tumor sampling.
* 13. Previous allogeneic bone marrow transplantation or solid organ transplantation.
* 14. Receipt of systemic anti-tumor therapy within 4 weeks prior to lymphodepletion conditioning, excluding the following situations:

  * Bridging therapy;
  * If prior treatment included nitrosourea or mitomycin chemotherapy, the interval between the end of chemotherapy and the expected start of lymphodepletion conditioning must be at least 6 weeks for enrollment;
  * If prior treatment included small-molecule targeted therapy, the interval between the end of treatment and the expected start of lymphodepletion conditioning must be at least 5 half-lives of the drug for enrollment.
* 15. Previous receipt of genetically modified or edited cell therapy products (excluding autologous immune cell therapy products without genetic modification or editing if more than 1 year has passed since cell infusion).
* 16. A history of hypersensitivity reactions to any component of the drugs intended for use in the study, including but not limited to autologous tumor-infiltrating lymphocytes (TILs), cyclophosphamide, fludarabine, interleukin-2 (IL-2), dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40, and antibiotics (β-lactam antibiotics, gentamicin).
* 17. Known history of mental illness, alcoholism, drug addiction, or substance abuse.
* 18. Previous grade 3 or higher adverse reactions to immunotherapy that failed to resolve to CTCAE grade 1 or below within 28 days; or any other disease or condition that could reasonably be suspected to contraindicate the use of investigational products, interfere with the interpretation of study results, or place the subject at high risk of treatment complications (including any other disease, metabolic disorder, abnormal physical examination finding, or abnormal laboratory test result).
* 19. Pregnant or lactating women; or women planning to become pregnant, lactate, or conceive within 1 year after cell infusion.
* 20. Receipt of other investigational products within 4 weeks prior to lymphodepletion conditioning, or planned participation in other investigational product studies during the study period.
* 21. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-12 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidience and severity of adverse events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection (GT201) in patients with relapsed/metastatic advanced solid tumor as measured by the incidience and severity of adverse events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China